CLINICAL TRIAL: NCT01260376
Title: Effect of Pharmacological Anti-lipolysis on FFA and VLDL-TG Metabolism Before and During Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Birgitte Nellemann, MD PhD student, University of Aarhus
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: M-20100221
Record Dates: First submitted 2010-12-13; First posted 2010-12-15 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Diabetes; Obesity
Keywords: VLDL-TG; Metabolism; Exercise; Free Fatty Acids
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Motor Activity | interventions — acipimox

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acipimox (Experimental): Tablet Acipimox 250 mg administered 4 times previous to and during the investigation day
  Interventions: Drug: Acipimox
- Placebo (No Intervention): Placebo tablets will be administered 4 times previous to and during the investigation day

INTERVENTIONS:
Drug: Acipimox — Tablet Acipimox 250 mg administered 4 times previous to and during the investigation day
  Arms: Acipimox

SUMMARY:
This study will investigate free fatty acid and VLDL-TG metabolism before and during exercise with and without pharmacological antilipolysis by the niacin antagonist Acipimox. Main focuses will be VLDL-TG and free fatty acid metabolism as well as expression of membrane proteins in fat- and muscle biopsies.

DETAILED DESCRIPTION:
Insulin resistance in liver and skeletal muscle is of central pathogenic significance in the development of type 2 diabetes. The molecular connections are unresolved but high levels of free fatty acids and triglyceride is probably involved. Diabetic subjects and to a lesser extent obese subjects have increased triglyceride levels, this could be due to an abnormal turnover of VLDL-TG. It is not yet investigated whether VLDL-TG kinetics changes during pharmacological antilipolysis. Using the aseptic ex-vivo labeling technique (developed in our laboratories) we will investigate this issue in sedentary healthy men. After a 3 hour basal period subjects will exercise on a bike for 60 minutes at 60% of VO2max. In both basal and exercise period one muscle and one fat biopsy will be obtained, further blood samples will be drawn to examine FFA and VLDL-TG metabolism etc..

This new knowledge will contribute to the understanding of metabolic disorders like type 2 diabetes and obesity.

ELIGIBILITY:
Inclusion Criteria:

- healthy, untrained males

Exclusion Criteria:

* medication
* history of malignancy, alcohol abuse or drug abuse
* participation in isotope trials in the last 6 months

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2011-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Effects of exercise and antilipolysis on FFA and VLDL-TG kinetics | 6 hour investigation day
  Healthy untrained men, investigated with pharmacological antilipolysis by Acipimox (Olbetam) and placebo on 2 occasions. Each day consists of 3 hour basal period and 90 minutes exercise on a bicycle at 60% of VO2-maximum. During the day glucose and lipid metabolism is investigated by glucose and VLDL tracer, as well as indirect calorimetrics. Cellular signaling is investigated by 2 muscle- and 2 fat biopsies each day.

CONTACTS AND LOCATIONS:
Overall Officials: Soren Nielsen, Dr. med., Principal Investigator — University Hospital of Aarhus
Locations (1):
- University Hospital of Aarhus, Norrebrogade, Aarhus, Aarhus, Denmark